CLINICAL TRIAL: NCT04667390
Title: Total Knee Arthroplasty Using an Active Robotic System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 199321
Record Dates: First submitted 2020-10-03; First posted 2020-12-14 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; the active robotic surgical system; robotic system in orthopedic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- total knee arthroplasty using the active robotic system (Active Comparator): total knee arthroplasty using the active robotic surgical system TSolution One TCAT, and system for planning TPlan
  Interventions: Other: total knee arthroplasty
- total knee arthroplasty using computer navigation (Active Comparator): Primary total knee arthroplasty using computer navigation and intraoperation control system
  Interventions: Other: total knee arthroplasty
- total knee arthroplasty using the standard manual tekhnik (Active Comparator): Primary total knee arthroplasty using the standard recommended set of instruments
  Interventions: Other: total knee arthroplasty

INTERVENTIONS:
Other: total knee arthroplasty — total knee arthroplasty

SUMMARY:
For the first time in Russia, it is planned to introduce and study primary knee arthroplasty using an active robotic system. The aim is to increase the efficiency of primary total knee arthroplasty using an active robotic surgical system. Traditional endoprosthetics of the knee joint (TKA) has now reached its maximum manufacturability and efficiency, but the accuracy of the performance depends on the skill and experience of the surgeon, as well as the efficiency of the cutting instrument (oscillator saw) when performing bone resection, the condition of the instrument and on the density of bone tissue fabric, which is highly variable. Modern RSS used in orthopedics include a robotic arm, robotic cutting devices with a computer navigation system, which are in active, semi-automatic or passive control mode. The main advantage of robotic systems is accurate preliminary planning using 3D modeling, use individual implant selection and virtual positioning.The active robotic surgical system TSolution-One allows participants to level the error in the positioning of the implant. The active robotic surgical system (ARSS) allows to correctly install the implant, which affects its service life, reduces the risks of postoperative complications, quickly returns to the usual way of life and forgets about the technical negative sensations and limitations that existed before the operation.It is planned to conduct an open-label retrospective and prospective clinical study in parallel observations.The study is planned to include 300 patients with osteoarthritis of the knee joint stage 3-4 (according to Kellgren-Lawrence). Investigators took three groups of patients, 100 patients each, and offered different options for total knee arthroplasty techniques.According to the research:-A clinical active robotic system for primary total knee arthroplasty will be introduced in Russia-There will be recommended indications and contraindications for this system in patients with gonarthrosis-The methodology of preoperative planning will be improved-The results of primary knee arthroplasty with an active robotic system will be evaluated in comparison with standard techniques and computer navigation-The methodology developed and improved in the dissertation will be introduced into the work of the clinical departments of traumatology, orthopedics and disaster surgery, studying the learning curve.

DETAILED DESCRIPTION:
Relevance: Robotic technologies were first introduced into medicine in the 1950s. The use of robotic systems in surgery begins with the use in neurosurgery. In 1985, the Programmable Universal Manipulation Arm (PUMA) 560 was introduced to perform CT-guided brain biopsy. In 1992, the Robodoc system (IBM) became the first orthopedic robotic system used in orthopedics for hip replacement, which subsequently improved the ability to automatically perform the stages of prosthetics. (Caspar system, Acrobot). Around the same time, the development of a robot for performing total knee arthroplasty began.

A distinctive feature of total knee arthroplasty (TKA) is the manufacturability of the stages and the high accuracy of surgical manipulations, which attracts the attention of many robotic surgical systems (RSS).

Traditional total knee arthroplasty (TKA) has now reached its maximum manufacturability and efficiency, but the accuracy of the performance depends on the skill and experience of the surgeon, as well as the accuracy of the cutting instrument (oscillator saw) when performing bone resection, the condition of the instrument and the density of the bone fabric, which is highly variable. The use of intramedullary guides during conventional surgery increases the risk of thromboembolic and cardiorespiratory complications. Computer navigation partially solves the problem of resection accuracy, infrared cameras read information from sensors and display a model with anatomical and kinematic features of the knee joint, which helps the surgeon to more accurately determine the level and direction of resection, but cannot ensure the accuracy of this manipulation and compliance with the preoperative plan.

Modern RSS used in orthopedics include a robotic arm, robotic cutting devices with a computer navigation system that operate in an active, semi-automatic, or passive control mode. The main advantage of robotic systems is accurate preoperative planning using 3D modeling, the possibility of individual selection of the implant and virtual positioning. Another advantage is the ability to accurately reproduce the preoperative plan during orthopedic surgery.

Today, active robotic surgical systems (ARSS) are used in clinical practice. ROBODOC / TSolution One. Robotic Surgical System (Curexo Technology, Fremont, Calif.), And Navio PFS (Blue Belt Technologies, Plymouth, Minnesota) Semi-Active Surgical Systems, OMNI Robotic System (OMNIlife Science, East Taunton, MA), RIO Robotic Arm Interactive Orthopedic System (Mako Surgical Corporation, Fort Lauderdale, Florida), ROSA Knee (Zimmer Zimmer Biomet, Montreal (Quebec), Canada).

The active robotic surgical system TSolution-One allows participants to level the error in the positioning of the implant. The accuracy of the filing is not affected by the manual skills of the surgeon, and does not depend on the density of bone tissue. Significant advantages of the system are: 1) precise preoperative breading; 2) rigid fixation of the limb, hip and tibia displacement sensors; 3) active autonomous milling without the participation of a surgeon; 4) accuracy of resection according to the preoperative plan; 5) rotation of the tibial component as in the preoperative plan; 6) no manual tools required; 7) postoperative control of the results of the operation. The active robotic surgical system (ARSS) allows participants to correctly install the implant, which affects its service life, reduces the risks of postoperative complications, the patient quickly returns to his usual way of life and forgets about those negative feelings and limitations that were before the operation.

The novelty of the proposed topic: For the first time in Russia, it is planned to introduce and study total knee arthroplasty using an active robotic system. Apply the use of a 3D patient model and the creation of an individual personalized preoperative plan using a robotic system for knee arthroplasty.

Aim and objectives of the research:

aim: To increase the efficiency of primary total knee arthroplasty using an active robotic surgical system.

objectives:

1. To study the possibilities of an active robotic system for primary arthroplasty of the knee joint, to determine indications and contraindications for use in endoprosthetics of the knee joint in patients with primary arthrosis.
2. To evaluate the technique of preoperative planning for total knee arthroplasty using an active robotic system in patients with arthrosis.
3. To work out the technique of total knee arthroplasty using an active robotic system, compare with computer navigation and the traditional method.
4. To evaluate the results of total knee arthroplasty using an active robotic system in comparison with the use of standard techniques and computer navigation.
5. Examine complications
6. Determine the place of the active robotic surgical unit in the total knee arthroplasty system.

Type of new research: an open-label, retrospective and prospective observational clinical study in parallel groups.

Research object and number of observations: the study is planned to include 300 patients with osteoarthritis of the knee joint of stage 3-4 (according to Kellgren-Lawrence).

Methods of the research:

1. General clinical examination of patients (collection of complaints, examination, assessment of physical findings and local status);
2. Assessment of the range of motion in the knee joint before and after surgery;
3. Performing X-ray images and CT of the knee joint before and after surgery, with the determination of the angles: LDFA, MPTA, Q, MAD;
4. Preoperative 3D planning on the TPLAN workstation;
5. Surgical treatment. 1) Primary total knee arthroplasty using the active robotic surgical system TSolution One, TCAT 2) Primary total knee arthroplasty using computer navigation 3) Primary total knee arthroplasty using the standard recommended set of instruments.
6. Evaluation of patient treatment results according to scales: VAS, KSS, OKS, WOMAC, SF-36, ASA, FJS-12, Spielberger test.
7. Methods of statistical processing of the material: statistical processing of data is planned to be carried out on a personal computer using Excel software packages and using standard methods of variation statistics using SPSS 16 statistical software packages.

Estimated research result:

1. For the first time in Russia, an active robotic system for primary total knee arthroplasty will be introduced into clinical practice.
2. Indications and contraindications for the use of this system in patients with gonarthrosis will be determined.
3. The methodology of preoperative planning will be improved.
4. The results of primary total knee arthroplasty using an active robotic system will be evaluated in comparison with the use of standard techniques and computer navigation.
5. The methodology developed and improved in the dissertation will be introduced into the work of the clinical bases of the Department of Traumatology, Orthopedics and Disaster Surgery, the study of the learning curve.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written informed consent of the patient to participate in the study;
2. Patients with stage 3-4 osteoarthritis of the knee joint (according to Kellgren-Lawrence.).
3. Men and women from 45 to 90 years old.
4. Pain in the knee joint above 3 points according to VAS
5. Opportunity for observations during the entire study period (12 months);
6. Mental adequacy, ability, willingness to cooperate and to fulfill the doctor's recommendations.

Exclusion Criteria:

1. Refusal of the patient from surgical treatment;
2. Presence of contraindications to surgical treatment;
3. Severe forms of diabetes mellitus (glycosylated hemoglobin> 9%);
4. Diseases of the blood (thrombopenia, thrombocytopenia, anemia with Hb <90 g / l);
5. The patient's unwillingness to conscious cooperation.
6. Refusal of the patient to participate in the study;
7. Non-compliance with the hospital regimen, according to the order of the Ministry of Health and Social Development of Russia dated 01.08.07, No. 514;
8. The impossibility of observing the patient within the control period after the operation.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Implant position assessment | 2 months after surgery
  CT scanning; these diagnostic methods assess the position of the implant, analysis of deformation, assessment of the angles in the knee joint ( LDFA, MPTA, MA, these diagnostic methods assess the position of the implant, analysis of deformation, assessment of the angles in the knee joint, analyze the rotation of implant).
Implant position assessment | 6 months after surgery
  CT scanning
Implant position assessment | 12 months after surgery
  CT scanning

OTHER OUTCOMES:
Quality of life and knee function assessment | 2,6,12 months after surgery
  Knee Society Score(KSS score), which combines subjective and objective information and separates the knee score (pain, stability, range of motion etc.) from the functional score of the patient (ability to walk, go up and down stairs).
Quality of life assessment ( joint awareness after surgery) | 2,6,12 months after surgery
  FJS-12, measures the clinical outcomes focusing on joint awareness after surgery
Spielberger test | 2,6,12 months after surgery
  Given these characteristics, test anxiety can be viewed as a situation-specific personality trait
Overall health score assessment | 2,6,12 months after surgery
  ASA score
Quality of life assessment (mental, physical assessment) | 2,6,12 months after surgery
  SF-36 score The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Quality of life assessment (the condition of patients) | 2,6,12 months after surgery
  WOMAC score is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints
Pain assessment | 2,6,12 months after surgery
  Visual Analog Score for pain (VAS)-dynamics pain assessment
Quality of life assessment (an individual's activities of daily living ) | 2,6,12 months after surgery
  OKS score The OKS is a patient reported outcome measure that consists of 12 questions about an individual's activities of daily living and how they have been affected by pain over the preceding four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Gritsyuk, PhD, Study Chair — First MSMU( I.M.Sechenov).The Department of Traumatology,Orthopedics
Locations (1):
- university clinical hospital № 1I.M.Sechenov First Moscow State Medical University. The Department of Traumatology, Orthopedics and Disaster Surgery, Moscow, Russia

REFERENCES:
- [Background] LYCHAGIN A.V.1, a, GRITSYUK A.A.1, b, RUKIN Y.A.1, c, ELIZAROV M.P.1, d, THE HISTORY OF THE DEVELOPMENT OF ROBOTICS IN SURGERY AND ORTHOPEDICS (LITERATURE REVIEW). 2020; 1 (39)2020: 10.17238/issn2226-2016.2020.1.13-19
- [Background] LYCHAGIN A.V. 1, a, RUKIN Y.A. 1, b, GRITSYUK A.A. 1, c, ELIZAROV M.P. 1, d, FIRST EXPERIENCE OF USING AN ACTIVE ROBOTIC SURGICAL SYSTEM IN TOTAL KNEE ARTHROPLASTY. 2019; 4 (38) 2019: 10.17238/issn2226-2016.2019.4.27-33